CLINICAL TRIAL: NCT06104527
Title: The Effect of Standard or Higher Protein Feeding on Indicator Amino Acid Oxidation in ICU Patients
Brief Title: Indicator Amino Acid Oxidation in ICU Patients
Acronym: IAAO-IC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NL84098.000.23
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; Muscle Wasting
Keywords: Dietary Protein; Enteral Nutrition
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.3 g/kg/day followed by 2.0 g/kg/day (Other): Patients in this arm will, on their first test day, receive enteral nutrition containing 1.3 grams of protein per kg of body weight per day followed by 2.0 grams of protein per kg of body weight per day on their second test day.
  Interventions: Combination Product: Standard protein enteral nutrition with enteral tracer; Combination Product: High protein enteral nutrition with enteral tracer
- 2.0 g/kg/day followed by 1.3 g/kg/day (Other): Patients in this arm will, on their first test day, receive enteral nutrition containing 2.0 grams of protein per kg of body weight per day followed by 1.3 grams of protein per kg of body weight per day on their second test day.
  Interventions: Combination Product: Standard protein enteral nutrition with enteral tracer; Combination Product: High protein enteral nutrition with enteral tracer

INTERVENTIONS:
Combination Product: Standard protein enteral nutrition with enteral tracer — Enteral nutrition with standard (1.3 g/kg/d) protein provision, given via a nasogastric tube. An oral L-[1-13C]-phenylalanine tracer is given as co-intervention. Use of an enterally given tracer is necessary to determine indicator amino acid oxidation.
Combination Product: High protein enteral nutrition with enteral tracer — Enteral nutrition with high (2.0 g/kg/d) protein provision, given via a nasogastric tube. An oral L-[1-13C]-phenylalanine tracer is given as co-intervention. Use of an enterally given tracer is necessary to determine indicator amino acid oxidation.

SUMMARY:
This study will use the indicator amino acid oxidation technique (IAAO) to determine protein oxidation of ICU patients at two protein intakes: 1.3 g/kg/d versus 2.0 g/kg/d.

DETAILED DESCRIPTION:
Rationale:

While protein administration guidelines for critical care are available from international organizations such as ASPEN and ESPEN, they vary greatly in their recommended dose and are based on relatively low-quality evidence. The Indicator Amino Acid Oxidation (IAAO) technique has been developed as a more practical and non-invasive tool to assess protein metabolism that can be used in vulnerable populations. Application of the IAAO technique in patients admitted to the Intensive Care Unit (ICU) could provide an alternative to better investigate optimal protein feeding during critical illness.

Objective:

To assess the effect of enteral feeding with higher protein content compared to standard protein content on indicator amino acid oxidation in ICU patients.

Study design:

Randomized, counterbalanced, cross-over trial.

Study population:

Adult patients with an unplanned admission to the ICU, who are mechanically ventilated and have an indication for prolonged enteral nutrition.

Intervention:

Subjects will undergo two test days in randomized order during which they receive either enteral feeding according to a standard protein dose (1.3 g/kg/d) or a higher protein dose (2.0 g/kg/d). Continuous feeding of L-[1-13C]-phenylalanine combined with breath, urine and blood samples will be applied to assess indicator amino acid oxidation.

Main study parameters/endpoints:

The primary endpoint is indicator amino acid oxidation after enteral feeding with a standard or higher protein content, determined using the Indicator Amino Acid Oxidation (IAAO) method by measuring 13CO2 enrichment in expired breath and enrichment of L-[1-13C]-phenylalanine in plasma and urine.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The overall risk of the study is negligible. The current study compares the effect of two nutritional compositions, that fall within the recommendations of international guidelines on ICU nutrition, on protein metabolism following ICU admission. To avoid overfeeding in the early phase of critical illness, both in terms of calories and protein, full enteral nutrition is provided after three days of gradual increase of intake (i.e., 25-50-75% of targeted intake, on days 1-2-3 respectively). Sampling of breath, urine, feces and plasma does not bring additional risks for this population. Our department has an extensive background in amino acid stable isotope methodology, assessment of 13CO2 enrichment in expired breath samples, and assessment of carbon dioxide production by indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Unplanned admission to the ICU
* Mechanically ventilated
* Start of enteral nutrition within 2 days of intubation
* ≥ 3 days on enteral nutrition
* Expected remaining ICU stay on mechanical ventilation of ≥ 2 days

Exclusion Criteria:

* Contra-indication for enteral nutrition at the discretion of the treating physician
* Feeding intolerance during incremental feeding protocol
* Moribund or withholding of treatment
* On extracorporeal membrane oxygenation (ECMO)
* Presence of chest drains, pneumothorax, tracheoesophageal fistula or subcutaneous emphysema
* Kidney failure AND a "no dialysis"-code on admission
* Hepatic encephalopathy (West Haven criteria 3-4)
* BMI < 18 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Indicator amino acid oxidation | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission.
  Indicator amino acid oxidation expressed as µmol/kg/h

SECONDARY OUTCOMES:
13CO2 excretion in breath (F13CO2) | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected before start of tracer and at end of tracer protocol.
  Collected using breath samples; measured using gas chromatography-mass spectrometry (Agilent G1530N/G2589A, Little Falls, USA)
Enrichments of plasma L-[1-13C]-phenylalanine | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected before start of tracer and at end of tracer protocol.
  Collected via in situ arterial catheter; measured using gas chromatography-mass spectrometry (Agilent G1530N/G2589A, Little Falls, USA)
Enrichments of urine L-[1-13C]-phenylalanine | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected before start of tracer and at end of tracer protocol.
  Collected via indwelling urinary catheter; measured using gas chromatography-mass spectrometry (Agilent G1530N/G2589A, Little Falls, USA)
Concentration of plasma phenylalanine | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected before start of tracer and at end of tracer protocol.
  Collected via in situ arterial catheter; analyzed using high performance liquid chromatography
Fecal output and fecal protein content | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected from start of intervention until end of intervention & tracer protocol.
  Collected via in situ fecal collection bag; protein content in fecal samples will be measured using Dumas method (Variomax CN-analyser)
Enrichment of breath 13CO2 | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected before start of tracer and at end of tracer protocol.
  Collected using breath samples; measured using gas chromatography-mass spectrometry (Agilent G1530N/G2589A, Little Falls, USA)
CO2 production | Collected at standard vs higher protein administration, on test day 1 and 2 (depending on randomisation order), during the first week of ICU admission. Per test day: collected 2 hours after start of tracer protocol.
  Measured using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Ph.D., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study data can be made available upon reasonable request, which will be considered by the project investigators (Drs. Julia Bels, Dr. Jorn Trommelen) and the Principal Investigator (Prof. Dr. Luc van Loon). A request for data-sharing together with a developed study protocol are prerequisites for consideration.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code